CLINICAL TRIAL: NCT06222398
Title: The Observation of Exoskeleton Use With In Home Functional Activities
Brief Title: Exoskeleton Use With In Home Functional Activities
Status: Terminated | Type: Observational
Why Stopped: We have finished all data collection for phase I and are not ready to start phase II
Sponsor: A.T. Still University of Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-196
Record Dates: First submitted 2023-12-18; First posted 2024-01-24 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-10

CONDITIONS: Paraplegia
MeSH Terms: conditions — Paraplegia | interventions — Exoskeleton Device

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Exoskeleton Users: This study includes patients who are current exoskeleton users. Exoskeleton users will engage in normal activities of daily living (ADLs) that they currently perform at wheelchair level while using the exoskeleton. Researchers will observe the ADLs the exoskeleton users are and are not able to complete while using their exoskeleton.
  Interventions: Device: Exoskeleton

INTERVENTIONS:
Device: Exoskeleton — The study will include one group of patients who are current exoskeleton users.

SUMMARY:
The purpose of this study is to observe current exoskeleton users in their home environment to determine the activities of daily living (ADLs) they are able to complete, and to identify the minor adaptations to the home environment that will improve the exoskeleton user's potential for increased independence. This is a pilot study to fine-tune the methods and to determine the feasibility of doing this study on a larger scale.

DETAILED DESCRIPTION:
The exoskeleton is a wearable robotic device that provides the ability to walk to those with spinal cord injury, or other neurological injuries who have lost their ability to walk and are wheelchair dependent. There are multiple health benefits to regaining the ability to adopt a standing posture, even for brief periods of time, including issues that are common with chronic wheelchair use such as pressure ulcers, bowel and bladder disorders, spasticity, and pain. Although there is a large amount of literature regarding people walking with the assistance of an exoskeleton, there is a dearth in the literature regarding use of an exoskeleton to complete normal activities of daily living (ADL) in the home environment. To date, no studies have been done assessing what the patient can do in their home environment while wearing the exoskeleton. The information that exists on the topic has been obtained primarily through interviews and surveys asking the patient to contemplate how to improve the exoskeleton, but patients have not been asked to complete ADLs wearing the exoskeleton, and their ability to do ADLs while using the exoskeleton has not been observed. As the ability to complete ADLs in standing would increase the usability of the exoskeleton, which would allow patients to wear them more frequently, and potentially for longer periods of time, this is a critical research gap. There is potential for physiological and psychological benefit to exoskeleton users with this increased use. It is possible that minor alterations in their environment could provide the opportunity for exoskeleton users to be independent, or nearly independent in some ADLs if their environment is set up for them. To determine these two points further research is indicated.

Specifically, for this study, patients who currently wear an exoskeleton will be observed in their home environment to determine the activities of daily living (ADLs) they are able to complete, and to identify the minor adaptations to the home environment that will improve the exoskeleton user's potential for increased independence. There will be one home visit where the environment for the patient will be adjusted as necessary (e.g. put necessary items on the counter or vanity so the patient can make a sandwich standing at the counter, or brush their teeth standing at the vanity). This minor adaptation provides easier access to items associated with activities of daily living. During this first visit, patients will complete several outcomes measures. The same outcome measures will be completed remotely, by phone or video call, by patients again at 1, 3, 6, 9, and 12 months post-initial home visit to determine if patients experience any change in the outcome measures (pain, quality of life, self-perception of task performance).

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* English speaking
* Trained and approved/credentialed by exoskeleton manufacturer to use the device independently according to FDA approved activities

Exclusion Criteria:

* Does not speak English
* <18 years of age
* Does not clearly meet inclusion criteria
* Has not been cleared by manufacturer for independent exoskeleton use

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population for this study is current exoskeleton users.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2024-02-10 (Actual); Primary Completion 2025-12-28 (Actual); Study Completion 2025-12-28 (Actual)

PRIMARY OUTCOMES:
Reintegration to Normal Living Index - Modified for Exoskeleton | baseline results will be collected same day as the home visit, same assessment will be repeated virtually at 1, 3, 6, 9, and 12 months
  Assesses quantitatively the degree to which individuals who have experienced traumatic or incapacitating illness achieve reintegration into normal social activities. This assessment has been modified from wheelchair level to exoskeleton level. The Reintegration to Normal Living Index has 9 Likert-style items. Each item is accompanied by verbal label choices with phrases reflecting how important the situation described is to the patient as it relates to using the exoskeleton. It allows the patients to determine the extent to which the statement in question applies to their specific situation.
Brief Pain Inventory (BPI) | baseline results will be collected same day as the home visit, same assessment will be repeated virtually at 1, 3, 6, 9, and 12 months
  The BPI allows patients to rate the severity of their pain and the degree to which their pain interferes with common dimensions of feeling and function.
  A higher score on the BPI indicates more severe pain. Scores can range from 0-10. The BPI scale defines pain as follows: Worst Pain Score: 1 - 4 = Mild Pain. Worst Pain Score: 5 - 6 = Moderate Pain. Worst Pain Score: 7 - 10 = Severe Pain.
Canadian Occupational Performance Measure (COPM) | baseline results will be collected same day as the home visit, same assessment will be repeated virtually at 1, 3, 6, 9, and 12 months
  The COPM assesses an individual's perceived occupational performance in the areas of self-care, productivity, and leisure.
  The COPM identifies 5 functional tasks the patient wants to improve, and rates their performance and satisfaction in their performance. Tasks are scored on a 1-10 scale (1-low; 10-high) for each item, then averaged over the 5 areas for an overall score. A higher score indicates better performance.

SECONDARY OUTCOMES:
Journal Entries | check journal monthly up to 12 months
  Participants will keep a daily journal/log for at least one month to keep track of how often they use the exoskeleton to do daily tasks, and to track their thoughts about using the exoskeleton in this way

CONTACTS AND LOCATIONS:
Overall Officials: Sue Dahl-Popolizio, DBH, Principal Investigator — A. T. Still University
Locations (1):
- A. T. Still University, Mesa, Arizona, United States

IPD SHARING:
Plan to Share IPD: No